CLINICAL TRIAL: NCT03879525
Title: Anxiety and Depression in Epilepsy: Assessing Outcomes Using the Electronic Medical Record (EMR)
Brief Title: EMR Outcomes: Anxiety and Depression in Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00056740
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-09

CONDITIONS: Quality of Life; Anxiety; Depression; Epilepsy
Keywords: Electronic medical record; EMR; Patient Outcomes
MeSH Terms: conditions — Anxiety Disorders; Depression; Epilepsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome group assignment will not be blinded to the primary investigator or primary study coordinator, as it will be necessary for these individuals to know outcome assessment allocation in order for outcome collection to occur. When possible, outcome group assignment will not be shared with the epilepsy provider managing the participant, in an effort to reduce any potential bias in retention that could be introduced by the provider in clinical interactions with the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMR Group (Experimental): Participants assigned to this arm will complete the questionnaires in the EMR using the EMR-based-interventional method.
  Interventions: Other: EMR-based-interventional method
- Phone Group (Active Comparator): Participants assigned to this arm will complete the questionnaires via the Phone using the Telephone-based-standard method.
  Interventions: Other: Telephone-based-standard method

INTERVENTIONS:
Other: EMR-based-interventional method — Questionnaire delivery method. Participants will complete standard care anxiety and depression screening and quality of life assessment directly into the patient entered section of the EMR, administered on arrival in the clinic.
  Arms: EMR Group
Other: Telephone-based-standard method — Questionnaires delivered via phone. Participants will complete standard care anxiety and depression screening and quality of life assessment via phone. Standard delivery method.
  Arms: Phone Group

SUMMARY:
The purpose of this research is to find out how people with epilepsy and possible symptoms of anxiety or depression are doing for 6 months after a regular epilepsy clinic visit. Participants in this study will complete questionnaires either by phone or via the patient portal.

DETAILED DESCRIPTION:
This is a study among N=30 individuals with epilepsy and high or borderline anxiety or depression symptoms receiving usual care at the Wake Forest Comprehensive Epilepsy Center. Participants are randomized to one of two outcome assessment methods [Electronic Medical Record (EMR)-based-interventional method vs. telephone-based-standard method] for collecting quality of life, anxiety and depression outcomes at 3 and 6 months, under usual care management.

The primary aim of the study is to assess feasibility of EMR-based outcome assessment by measuring 6-month retention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Completed electronic questionnaires independently in clinic
* Epilepsy diagnosis (clinician impression or EEG-based)
* Borderline or high anxiety or depression symptoms at baseline
* GAD-7 score > 7 (anxiety)
* NDDI-E score > 13 (depression)

Exclusion Criteria:

* Passive suicidal ideation (NDDI-E item 4 score of 3 or 4)
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi M. Munger Clary, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Will consider requests if received.

RESULTS

PARTICIPANT FLOW:
Groups:
- EMR Group: Participants assigned to this arm will complete the questionnaires in the Electronic Medical Record (EMR) using the EMR-based-interventional method.
  EMR-based-interventional method: Questionnaire delivery method. Participants will complete standard care anxiety and depression screening and quality of life assessment directly into the patient entered section of the EMR, administered on arrival in the clinic.
Period: Overall Study
Arm/Group | EMR Group | Phone Group
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EMR Group | Phone Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.4) | 42.5 (12.7) | 42.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 11 | 12 | 23
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Retained in the Study in the EMR Arm
Description: Retention is defined as the percentage of participants in the study who complete the 6 month outcome instruments in the EMR
Time Frame: 6 months
Population: This outcome pertains only to EMR group; phone group is analyzed in separate outcome.
Measure: Number; unit: percentage of participants
Arm/Group | EMR Group
Number analyzed (Participants) | 15
percentage of participants | 67

2. Secondary Outcome: Percentage of Participants Retained in the Study in the Phone Arm
Description: Retention is defined as the percentage of participants in the study who complete the 6 month outcome instruments via phone
Time Frame: 6 months
Population: This outcome pertains only to the phone group; EMR group was analyzed in a different outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Phone Group
Number analyzed (Participants) | 15
percentage of participants | 100

3. Secondary Outcome: Quality of Life in Epilepsy-10 (QOLIE-10)
Description: QOLIE-10 is A brief questionnaire (10-items) to screen for quality of life in epilepsy. Total Score 0-100. Higher scores denotes worse outcomes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMR Group | Phone Group
Number analyzed (Participants) | 15 | 15
score on a scale | 53.3 (16.6) | 60.5 (18.6)

4. Secondary Outcome: Quality of Life in Epilepsy-10 (QOLIE-10)
Description: as for outcome 3
Time Frame: 3 Months
Population: 5 individuals in EMR arm did not return the 3 month outcome assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMR Group | Phone Group
Number analyzed (Participants) | 10 | 15
score on a scale | 61.0 (18.6) | 57.3 (15.7)

5. Secondary Outcome: Quality of Life in Epilepsy-10 (QOLIE-10)
Description: as for outcome 3
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMR Group | Phone Group
Number analyzed (Participants) | 15 | 15
score on a scale | 57.6 (20.3) | 62.6 (16.7)

6. Secondary Outcome: Generalized Anxiety Disorder 7-item (GAD-7) Scale
Description: Anxiety scale. Total Score 0-28. Higher scores denotes worse outcomes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMR Group | Phone Group
Number analyzed (Participants) | 15 | 15
score on a scale | 10.5 (5.3) | 10.5 (3.8)

7. Secondary Outcome: Generalized Anxiety Disorder 7-item (GAD-7) Scale
Description: Anxiety scale. Total Score 0-28. Higher scores denotes worse outcomes.
Time Frame: 3 Months
Population: 5 individuals in EMR arm did not return the 3 month outcome assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMR Group | Phone Group
Number analyzed (Participants) | 10 | 15
score on a scale | 6.0 (3.0) | 10.2 (4.2)

8. Secondary Outcome: Generalized Anxiety Disorder 7-item (GAD-7) Scale
Description: Anxiety scale. Total Score 0-28. Higher scores denotes worse outcomes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMR Group | Phone Group
Number analyzed (Participants) | 15 | 15
score on a scale | 7.7 (5.4) | 8.5 (5.0)

9. Secondary Outcome: Neurological Disorders Depression Inventory (NDDI-E)
Description: The NDDI-E is a 6-item questionnaire validated to screen for depression in people with epilepsy. Total Score 4-24. Higher scores denotes worse outcomes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMR Group | Phone Group
Number analyzed (Participants) | 15 | 15
score on a scale | 15.4 (2.8) | 15.3 (3.4)

10. Secondary Outcome: Neurological Disorders Depression Inventory (NDDI-E)
Description: as for outcome 9
Time Frame: 3 Months
Population: 5 individuals in EMR arm did not return the 3 month outcome assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMR Group | Phone Group
Number analyzed (Participants) | 10 | 15
score on a scale | 15.4 (3.1) | 15.0 (2.6)

11. Secondary Outcome: Neurological Disorders Depression Inventory (NDDI-E)
Description: as for outcome 9
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMR Group | Phone Group
Number analyzed (Participants) | 15 | 15
score on a scale | 14.7 (3.9) | 13.8 (3.4)

12. Other Pre Specified Outcome: Semi-Structured Interviews
Description: Optional semi-structured interviews to assess patient-level barriers and facilitators to successfully implementing a collaborative care model of mental health care. Data will be analyzed via an inductive thematic analysis approach.
Time Frame: 13 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through 6 month follow up
Arm/Group | EMR Group | Phone Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMR Group (N=15) | Phone Group (N=15)
status epilepticus (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT03879525/Prot_SAP_001.pdf
  • Informed Consent Form (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT03879525/ICF_000.pdf